CLINICAL TRIAL: NCT04711837
Title: A Multicenter, Randomized, Double-blinded, Propofol-controlled, Phase 3 Clinical Study to Evaluate the Efficacy and Safety of HSK3486 Injectable Emulsion for Induction of General Anesthesia in Adults Undergoing Elective Surgery.
Brief Title: Efficacy and Safety of HSK3486 Compared to Propofol in Induction of General Anesthesia in Adults Having Elective Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco-USA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK3486-304
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Anesthesia
Keywords: Anesthesia; Elective surgery; Propofol
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): HSK3486 for induction of general anesthesia.
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): Propofol for induction of general anesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — HSK3486 for induction of general anesthesia.
  Arms: HSK3486
Drug: Propofol — Propofol for induction of general anesthesia.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
This is a multicenter, randomized, double-blinded, propofol-controlled, Phase 3 clinical study to evaluate the efficacy and safety of HSK3486 for induction of general anesthesia in adults undergoing elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing elective surgery (nonemergency, noncardiothoracic, and nonintracranial surgery anticipated to last at least 1 hour ).
* Males or females, aged ≥18 years old, with American Society of Anesthesiologists Physical Status (ASA PS) I to IV.
* Body mass index (BMI) ≥18 kg/m2.
* For all females of childbearing potential, negative pregnancy test at screening and baseline. Additionally, females of childbearing potential must agree to use birth control (such as condom, intrauterine device [IUD], abstinence) from the time of consent until 30 days post study drug administration.
* Capable of understanding the procedures and methods of this study, willing to sign an Informed Consent Form, and to complete this study in strict compliance with the study protocol.

Exclusion Criteria:

* Contraindications to deep sedation/general anesthesia or a history of adverse reaction to sedation/general anesthesia.
* Known to be allergic to eggs, soy products, opioids and their antidotes, or propofol; subject having contraindications to propofol, opioids, and their antidotes.
* Medical condition or evidence of increased sedation/general anesthesia risk.
* Management risks of respiratory tract and judged by the investigator to be unsuitable for inclusion in the study.
* Any medication that has the potential to interact synergistically with propofol or HSK3486, including but not limited to all sedatives and hypnotics.
* Laboratory parameters significantly out of range at screening.
* Female subjects with a positive pregnancy test (serum or urine) at screening or baseline; lactating subjects; any subject planning to get pregnant within 1 month after the study (including the male subject's partner).
* Judged by the investigator to have any other factors that make the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Daley, MD, Study Director — Haisco-USA Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - Arizona Research Center, Phoenix, Arizona
  - Lotus Clinical Research, LLC, Pasadena, California
  - Phoenix Clinical Research, LLC, Tamarac, Florida
  - The University of Chicago Medicine, Chicago, Illinois
  - New York City Heath and Hospitals, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - UNC Health Care System, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The Ohio State University Research Foundation, Columbus, Ohio
  - HD Research, Bellaire, Texas
  - Plano Surgical Hospital, Plano, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - JBR Clinical Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HSK3486 | Propofol
Started | 170 | 85
Completed | 168 | 83
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HSK3486 | Propofol | Total
Number analyzed (Participants) | 168 | 83 | 251
Age, Customized [Count of Participants; unit: Participants]
  Age Group (Years): ≥65 | 27 | 14 | 41
  Age Group (Years): <65 | 141 | 69 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 57 | 176
  Male | 49 | 26 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 23 | 68
  Not Hispanic or Latino | 118 | 58 | 176
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 12 | 48
  White | 121 | 71 | 192
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Anesthesia Induction
Description: The primary outcome of interest was the success rate of anesthesia induction, defined by the proportion of subjects with successful anesthesia. A subject was considered successful for anesthetic induction if the following conditions were met: induction success Modified Observer's Assessment of Awareness/Sedation Scale (MOAA/S ≤1) after administration of study drug and 1 or less top-up dose required without using any rescue drugs. Where Grade 0 is no response after trapezius squeeze, Grade 1 responds only after painful trapezius squeeze and Grade 5 is completely awake responds to name spoken in normal tone.
Time Frame: From start of drug administration to MOAA/S ≤1 (up to 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 168 | 83
Participants | 163 | 81

2. Secondary Outcome: Subjects' NRS Pain Score
Description: Injection-site pain is evaluated verbally during study drug administration using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worse imaginable pain). Subjects' NRS pain score at the time of study drug administration (Day 1) and recall of pain score in PACU.
Time Frame: Up to 8 hours
Population: Full Analysis Set (FAS): All randomized subjects who have received at least 1 dose of the study drug (HSK3486 or propofol).
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 168 | 83
Participants
  Proportion of NRS ≥ 1 pain score on Day 1: Proportion of NRS ≥1 and <4 pain score | 20 | 13
  Proportion of NRS ≥ 1 pain score on Day 1: Proportion of NRS ≥4 pain score | 10 | 51
  Proportion of NRS ≥ 1 pain score on Day 1: Proportion of NRS = 0 Pain score | 137 | 19
  Proportion of NRS ≥ 1 pain score on Day 1: Missing NRS | 1 | 0
  Proportion of NRS ≥ 1 pain Score in PACU: Proportion of NRS ≥1 and <4 pain score | 27 | 17
  Proportion of NRS ≥ 1 pain Score in PACU: Proportion of NRS ≥4 pain score | 19 | 39
  Proportion of NRS ≥ 1 pain Score in PACU: Proportion of NRS = 0 Pain score | 113 | 21
  Proportion of NRS ≥ 1 pain Score in PACU: Missing NRS | 9 | 6

3. Secondary Outcome: Proportion of Subjects With Successful Induction Who Maintain the Desired Depth of Anesthesia for General Elective Surgery, AND Without Significant Cardiac and Respiratory Depression.
Description: The proportion of subjects with successful induction who maintain the desired depth of anesthesia for general elective surgery, AND without significant cardiac and respiratory depression between the time of successful induction and 15 minutes post initiation of study drug administration, or up to the beginning of second tracheal intubation attempt if it is a difficult condition and not beyond 15 minutes post initiation of study drug administration.
Time Frame: 15 minutes from end of drug administration.
Population: Induction of General Anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 168 | 83
Participants
  Successful Induction | 163 | 81
  Failed Induction | 5 | 2

4. Secondary Outcome: Proportion of Subjects With Any Injection-site Pain on Numeric Rating Scale.
Description: The proportion of subjects with any injection-site pain at time of drug administration on the Numeric Rating Scale (NRS ≥1).
Time Frame: From start of drug administration to MOAA/S ≤1 (up to 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 167 | 83
Participants | 30 | 64

5. Secondary Outcome: Time to Successful Induction of General Anesthesia.
Description: Time from the end of the first administration of the study drug to MOAA/S ≤1.
Time Frame: From end of drug administration to MOAA/S ≤1 (up to 5 minutes)
Population: Time to successful induction of general anesthesia was defined as the time from the end of first administration of the study drug to the time when MOAA/S was ≤1.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 168 | 83
minutes | 0.75 [0.6167 to 0.9000] | 0.62 [0.5167 to 0.8000]

6. Other Pre Specified Outcome: Time to the Disappearance of Eyelash Reflex
Description: Time from the end of the first administration of the study drug to the disappearance of eyelash reflex.
Time Frame: From end of drug administration to disappearance of eyelash reflex (up to 5 minutes)
Population: Time to loss of eyelash reflex was defined as the time from the end of the first administration of the study drug to the time when eyelash reflex was lost.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 168 | 83
minutes | 0.92 [0.8333 to 1.0000] | 0.80 [0.7333 to 1.0000]

7. Other Pre Specified Outcome: Number of Participants That Failed to Meet Successful Induction of General Anesthesia
Description: Failed to meet successful induction of general anesthesia defined by the use of the Top-up Study Drug and Rescue/Remediation Drugs
Time Frame: From start of drug administration to MOAA/S ≤1 (up to 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 168 | 83
Participants | 5 | 2
Statistical Analysis 1: Comparison: HSK3486 vs Propofol; Test type: Non-Inferiority — Non-inferiority margin equals to -8%; Farrington-Manning method — Non-inferiority margin equals to -8%: 95% CI; (-5.4%, 4.2%); Risk Difference (RD) = -0.0057, 95% CI 2-sided [-0.054 to 0.042], Standard Error of Mean 0.0246

ADVERSE EVENTS:
Time Frame: Adverse event reporting begins from the time of informed consent and ends 30 days after the last dose of study drug.
Arm/Group | HSK3486 | Propofol
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/168 | 3/83
Other Adverse Events (participants affected / at risk) | 47/168 | 27/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSK3486 (N=168) | Propofol (N=83)
Pulmonary Embolism (Cardiac disorders) | 0 (0) | 1 (83)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 (0) | 1 (83)
Femur Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (83)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HSK3486 (N=168) | Propofol (N=83)
Hypotension (Vascular disorders) | 47 | 27
Nausea (Gastrointestinal disorders) | 46 | 27
Procedural Pain (Injury, poisoning and procedural complications) | 32 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT04711837/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT04711837/SAP_001.pdf